CLINICAL TRIAL: NCT04420897
Title: The Effect of Intraoperative Arterial Oxygen Pressures on Early Post-Operative Patient and Graft Survival in Living Donor Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bora Dinc, Assistant Professor Department of Anesthesiology and Reanimation, Akdeniz University
Other Study IDs: The effect of Pa02 in KT
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Kidney Transplant; Complications; Hyperoxia; Graft Dysfunction
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normoxy: PaO2 = 80-120 mm Hg: Data collection explained below: Arterial blood samples from all groups shall be taken after induction, 5 minutes after graft perfusion, and end of surgery in the intraoperative period, in the operating room. The duration of the intensive care unit (ICU), the duration of mechanical ventilation in intensive care, Whether or not to re-intubate, hospital stay, intraoperative and postoperative laboratory data, immunosuppression regimen, postoperative complications (surgical site infection, ischemic vascular conditions, complications from respiratory) and interventions will be included for the study analysis. The survival of the patients will be enrolled, and the relationship between the obtained data and survival will be investigated. For early-stage graft survival, postoperatively; Data such as renal replacement therapy, the total amount of urine levels, creatinine values, presence of delayed graft function will be recorded.
  Interventions: Procedure: Arterial blood gas samples
- Moderate hyperoxemia: PaO2 =120-200 mm Hg: Data collection explained below: Arterial blood samples from all groups shall be taken after induction, 5 minutes after graft perfusion, and end of surgery in the intraoperative period, in the operating room. The duration of the intensive care unit (ICU), the duration of mechanical ventilation in intensive care, Whether or not to re-intubate, hospital stay, intraoperative and postoperative laboratory data, immunosuppression regimen, postoperative complications (surgical site infection, ischemic vascular conditions, complications from respiratory) and interventions will be included for the study analysis. The survival of the patients will be enrolled, and the relationship between the obtained data and survival will be investigated. For early-stage graft survival, postoperatively; Data such as renal replacement therapy, the total amount of urine levels, creatinine values, presence of delayed graft function will be recorded.
  Interventions: Procedure: Arterial blood gas samples
- Severe hyperoxemia: PaO2 >200 mm Hg: Data collection explained below: Arterial blood samples from all groups shall be taken after induction, 5 minutes after graft perfusion, and end of surgery in the intraoperative period, in the operating room. The duration of the intensive care unit (ICU), the duration of mechanical ventilation in intensive care, Whether or not to re-intubate, hospital stay, intraoperative and postoperative laboratory data, immunosuppression regimen, postoperative complications (surgical site infection, ischemic vascular conditions, complications from respiratory) and interventions will be included for the study analysis. The survival of the patients will be enrolled, and the relationship between the obtained data and survival will be investigated. For early-stage graft survival, postoperatively; Data such as renal replacement therapy, the total amount of urine levels, creatinine values, presence of delayed graft function will be recorded.
  Interventions: Procedure: Arterial blood gas samples

INTERVENTIONS:
Procedure: Arterial blood gas samples — Blood gases taken during the operation will be analyzed retrospectively. Whether these results have an effect on graft survival will be examined by reaching their records in the postoperative period.

SUMMARY:
We evaluated the prognostic role of the intraoperative arterial oxygen partial pressures (PaO2) on postoperative patient and graft survival in living donor kidney transplantations.

DETAILED DESCRIPTION:
Undoubtedly, one of the most important elements of life on earth is oxygen. Aerobic organisms adapted to the 20.8% oxygen ratio in the atmosphere have survived even lower than this concentration by developing various defense mechanisms. The real question is whether high levels of oxygen in the blood, which are administered iatrogenically, leads to tissue destruction.

Reactive Oxygen Species (ROS), which is a result of hyperoxia and may be useful even at low levels, may cause tissue loss due to oxidative stress, also called oxygen-free radicals. ROS, whose toxicity is very destructive with its accumulation, may cause damage to macromolecular structures such as lipids, protein, mitochondrial and nuclear DNA. On the organs of the exposed oxidative stress; For lung, asthma, chronic obstructive pulmonary disease (COPD), acute respiratory distress syndrome (ARDS), cardiovascular system, ischemic heart disease (IHD), hypertension, shock, heart failure, while kidney failure and glomerulonephritis can cause unwanted complications.

The kidneys get for circulation, only 20% of the cardiac output. Since the arterial and venous (AV) structures in the kidneys are anatomically parallel to each other, the oxygen concentration in the renal vein may be relatively higher than the efferent arteriole and cortex because of the oxygen shunt. Thanks to this mechanism, in clinical situations where partial oxygen pressure (Pa02) is high, the oxygen concentration presented to the kidney tissues remains within a certain limit. In fact, AV shunt protects kidney tissue with a structural antioxidant mechanism. Thus, the increase in renal blood flow (RBF) will cause an increase in AV oxygen shunt in parallel, the blood coming to the kidneys participates in the systemic circulation without entering the renal microcirculation. It has been suggested that shunt occurs to protect from hyperoxia at the tissue level by decreasing blood volume in the kidneys. Oxidative stress, which is inevitable as a result, will increase tissue hypoxia paradoxically by increasing the oxygen consumption of the kidneys. It is stated that uremic toxin, especially indoxyl sulfate (IS) accumulation is the cause of the mentioned table. Apart from IS, phenyl sulfate and ρ-cresy sulfate make tubular cells susceptible by reducing glutathione levels. Thus, increased renal hypoxia, renal oxidative stress will result in renal inflammation and fibrosis.

According to recent studies, the antioxidant defense mechanism has been shown not only to be limited to AV shunt. But also the dynamic regulation of intrarenal oxygenation in RBF changes. However, mechanisms developed to prevent hyperoxia have made kidney tissue sensitive to hypoxia. The increase in AV oxygen shunt causes an increase in tissue hypoxia.

Although endogenous antioxidant mechanisms play a major role against free radicals, the postoperative effects of iatrogenic hyperoxia on transplanted kidney grafts and patient survival remain a subject to be investigated. That's why we aim to understand the impact of iatrogenic hyperoxia during the living donor kidney transplantation operations by retrospective data analyzing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had living donor kidney transplantation between January 2014 and June 2019 at Akdeniz University Faculty of Medicine Organ Transplant Center.

Exclusion Criteria:

* Patients with missing data
* Patients with a history of chronic heart failure or chronic respiratory disease (bronchial asthma, COPD).
* Presence of cadaveric donor kidney transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled only 1000 adult living donor kidney transplantations closed files started from 1st of January 2017 to 1st of November 2019. The study conducted at the Department of Anesthesiology and Critical Care with the Department of General and Visceral Surgery Medical Center. All recipient surgical procedure was carried out by the same specialized transplantation surgeons and anesthesiologists after a positive vote of the local ethics committee for transplantation. Recipients with a history of myocardial infarction, chronic respiratory disease (bronchial asthma, COPD) were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of arterial blood gases with normoxia | Postoperative first following month
  Approximately 1000 patients enrolled have living donor renal transplantation. After separation by study limitation of the accepted groups according to the PaO2 levels, graft functions and the patient's prognosis will be evaluated by enrolled data gained during the postoperative first month.
Assessment of arterial blood gases with Moderate hyperoxemia | Postoperative first following month
  Approximately 1000 patients enrolled have living donor renal transplantation. After separation by study limitation of the accepted groups according to the PaO2 levels, graft functions and the patient's prognosis will be evaluated by enrolled data gained during the postoperative first month.
Assessment of arterial blood gases with Severe hyperoxemia | Postoperative first following month
  Approximately 1000 patients enrolled have living donor renal transplantation. After separation by study limitation of the accepted groups according to the PaO2 levels, graft functions and the patient's prognosis will be evaluated by enrolled data gained during the postoperative first month.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Di̇nc, MD, Assist. Prof., Principal Investigator — Akdeniz University Medical Faculty
Locations (1):
- Akdeniz University Medical Faculty Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Dinc B, Yilmaz VT, Aycan IO, Kisaoglu A, Dandin O, Aydinli B, Hadimioglu N, Ertug Z. Effect of post-perfusion hyperoxemia on early graft function in renal transplant recipients: a retrospective observational cohort study. Ir J Med Sci. 2021 Nov;190(4):1539-1545. doi: 10.1007/s11845-020-02499-7. Epub 2021 Jan 4. PMID 33398714